CLINICAL TRIAL: NCT02315768
Title: A Phase Ib/II Study of Ibrutinib in Combination With GA101 - Obinutuzumab in Previously Untreated Chronic Lymphocytic Leukemia (CLL) Patients Over 65 Years of Age or With Comorbidities That Preclude the Use of Chemotherapy Based Treatment
Brief Title: Ibrutinib in Combination With GA101 (Obinutuzumab) in Previously Untreated Chronic Lymphocytic Leukemia (CLL) Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Principal Investigator, Thomas Kipps, Deputy Director, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 141106
Record Dates: First submitted 2014-10-30; First posted 2014-12-12 (Estimated); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Chronic Lymphocytic Leukemia; Ibrutinib; Obinutuzumab; Cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — obinutuzumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GA101+ibrutinib (Experimental): Ibrutinib 420 mg (140 mg capsules 3 times) orally once daily for up to 6 cycles.
  GA101 (Obinutuzumab) by Intravenous infusion for up to 6 cycles (28 day cycles) as follows:
  * Cycle 1, Day 1,100 mg GA101 obinutuzumab will be administered.
  * Cycle 1, Day 2, 900 mg of GA101 obinutuzumab will be administered.
  * Cycle 1, Days 8 and 15,1,000 mg of GA101 obinutuzumab will be administered.
  * Cycles 2-6, Day 1, 1,000 mg of GA101 obinutuzumab will be administered.
  Interventions: Drug: GA101; Drug: Ibrutinib

INTERVENTIONS:
Drug: GA101
  Other Names: Obinutuzumab
Drug: Ibrutinib
  Other Names: Imbruvica

SUMMARY:
The purpose of the study is to determine whether ibrutinib in combination with GA101 - Obinutuzumab might be useful for the treatment of CLL. This study will evaluate if ibrutinib in combination with GA101 - Obinutuzumab can reduce the amount of cancerous cells in body.

DETAILED DESCRIPTION:
This is an open label phase IB/II clinical trial designed to determine the safety and clinical activity of Ibrutinib in combination with GA101 - Obinutuzumab. Safety, tolerability and dose-limiting toxicities (DLTs) will be evaluated during the initial cycle of treatment (Cycle 1; Day 1-28) as part of the phase Ib of this study (safety run-in).

In the phase II the response rate will be determined in all subjects that have received treatment. The study will enroll 32 subjects previously untreated who have active disease requiring treatment (as defined by IWCLL 2008 criteria for initiation of therapy). The study will include a Screening Phase, a Treatment Phase, and a Follow-up Phase. The Screening Phase assessments will be performed within 28 days prior to treatment. The Treatment Phase will extend from first dose until completion of all planned cycles of treatment (#6) or study drug discontinuation.

All subjects will receive Ibrutinib 420 mg (3 x 140-mg capsules) orally once daily for up to 6 cycles. The treatment with Ibrutinib will continue after cycle 6 for the following 3 years until disease progression, unacceptable toxicity or other reason for treatment discontinuation.

Subjects will undergo response assessment two months after completion of the study treatment. The initial follow-up evaluations will be made (after the response assessment) every 3 months during 9 months and later every 6 months until initiation of new treatment for CLL, consent withdrawal or death. During the long-term follow-up phase, subjects will be followed for survival (PFS, TFS and OS). The long-term follow-up phase will continue until disease progression, death, loss to follow up, consent withdrawal, or study end, whichever occurs first.

An evaluation of the End of Study will be performed due to initiation of new treatment for CLL or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CLL
2. Indication for treatment as defined by the International Workshop on Chronic Lymphocytic Leukaemia (IWCLL) Guidelines
3. No previous treatment for CLL
4. Males and females 65 years of age and older. Subjects under 65 years of age that meet any of the following criteria:

   A. Documented refusal to be treated with chemotherapy agents B. Subjects that are not candidates for treatment with chemotherapy based on poor performance status (ECOG g>= 2), Cumulative Illness Rating Scale (CIRS score) >= 6 or creatinine clearance less than 70 mL/min
5. Adequate hematologic, hepatic, and renal function
6. Anticipated survival of at least 6 months
7. Effective contraception is required while receiving Ibrutinib in combination with GA101-Obinutuzumab. For women of childbearing potential and men, effective contraception is required while receiving GA101-Obinutuzumab and for 365 days (12 months) after the last dose of the study drug

Exclusion Criteria:

1. Pregnant or nursing women
2. Treatment with chemotherapy, monoclonal antibodies, or biological agents (e.g. lenalidomide) other than the investigational agents during the time of participation in this trial
3. Grade 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
4. Severe or debilitating pulmonary disease
5. Participation in any investigational drug study within 28 days prior to initiation of treatment within this protocol.
6. History of second malignancy, other than non-melanoma skin cancer or in situ carcinoma of the cervix or the breast, unless the tumor was successfully treated at least 2 years before trial entry and with no evidence of relapse or active cancer.
7. Active symptomatic fungal, bacterial and/or viral infection including evidence of infection with HIV, human T-cell leukemia virus 1 (HTLV-1) seropositive status.
8. Evidence of active acute or chronic Hepatitis B (HBV)
9. Evidence of active Hepatitis C (HCV): subjects with positive hepatitis C serology and positive HCV RNA test
10. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
11. Known hypersensitivity to any of the study drugs
12. Major surgery (within 4 weeks prior to the start of Cycle 1), except for procedures that are performed for diagnostic purposes
13. Vaccination with a live vaccine within 28 days of the initiation of treatment.
14. Concomitant use of warfarin or other Vitamin K antagonists
15. Requirement to receive treatment with a strong cytochrome P450 (CYP) 3A inhibitor
16. Chronic liver disease with hepatic impairment (Child-Pugh class B or C)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Kipps, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Castro JE, Lengerke-Diaz PA, Velez Lujan J, Choi MY, Moreno-Cortes EF, Forero JV, Garcia-Robledo JE, Jacobs C, McCarthy C, Heinen A, Amaya-Chanaga CI, Kipps TJ. Ibrutinib plus Obinutuzumab as Frontline Therapy for Chronic Lymphocytic Leukemia Is Associated with a Lower Rate of Infusion-Related Reactions and with Sustained Remissions after Ibrutinib Discontinuation: A Single-Arm, Open-Label, Phase 1b/2 Clinical Trial NCT0231576. Adv Hematol. 2022 Jan 22;2022:4450824. doi: 10.1155/2022/4450824. eCollection 2022. PMID 35103064

RESULTS

PARTICIPANT FLOW:
Groups:
- GA101+Ibrutinib: Ibrutinib 420 mg (140 mg capsules 3 times) orally once daily for up to 6 cycles.
  GA101 (Obinutuzumab) by Intravenous infusion for up to 6 cycles (28 day cycles) as follows:
  * Cycle 1, Day 1,100 mg GA101 obinutuzumab will be administered.
  * Cycle 1, Day 2, 900 mg of GA101 obinutuzumab will be administered.
  * Cycle 1, Days 8 and 15,1,000 mg of GA101 obinutuzumab will be administered.
  * Cycles 2-6, Day 1, 1,000 mg of GA101 obinutuzumab will be administered.
  GA101
  ibrutinib
Period: Overall Study
Arm/Group | GA101+Ibrutinib
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GA101+Ibrutinib
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Safety, Tolerability and Dose Limiting Toxicity (DLT) of Ibrutinib in Combination With Obinutuzumab
Description: Remission rate after discontinuation of Ibrutinib in patients with previously untreated CLL treated with Ibrutinib in combination with Obinutuzumab
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GA101+Ibrutinib
Number analyzed (Participants) | 32
Participants | 32

2. Primary Outcome: Overall Response Rate of Ibrutinib in Combination With Obinutuzumab
Description: Determine the overall response rate of Ibrutinib in combination with Obinutuzumab in previously untreated subjects with CLL. Overall response rate was based on the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2008 criteria.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GA101+Ibrutinib
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Time Frame: 3 years
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | GA101+Ibrutinib
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA101+Ibrutinib (N=32)
Fever/Sepsis (IRR) (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
SAE (General disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA101+Ibrutinib (N=32)
Abdominal cramping (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Albumin decreased (General disorders) | 1 (1)
Alkaline Phosphatasee Increase (Hepatobiliary disorders) | 2 (6)
ALT elevated (Hepatobiliary disorders) | 11 (19)
Anemia (Blood and lymphatic system disorders) | 6 (12)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
AST elevated (Hepatobiliary disorders) | 11 (16)
Atrial fibrillation (Cardiac disorders) | 3 (6)
Back and neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bleeding from auditory cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Hepatobiliary disorders) | 6 (16)
Brittle nails (Skin and subcutaneous tissue disorders) | 4 (4)
Bruising (Vascular disorders) | 7 (8)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Chronic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Creatinine increased (Renal and urinary disorders) | 5 (14)
Diarrhea (Gastrointestinal disorders) | 15 (23)
Dry Mouth (General disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Ear bleeding (Ear and labyrinth disorders) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 1 (1)
edema (Vascular disorders) | 2 (2)
Elevated AST (Hepatobiliary disorders) | 10 (12)
Elevated Bilirubin (Hepatobiliary disorders) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 5 (8)
Elevated Phosphorus (Renal and urinary disorders) | 1 (1)
Elevated uric acid (Renal and urinary disorders) | 1 (1)
Epistaxis (General disorders) | 3 (3)
Eye Infection (Eye disorders) | 1 (1)
Facial bruise (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 5 (7)
Fever (General disorders) | 9 (10)
Fever (General disorders) | 2 (3)
Finger Nail Fragility (Skin and subcutaneous tissue disorders) | 1 (1)
Flu-like symptoms (General disorders) | 2 (4)
Fragile Nails (Skin and subcutaneous tissue disorders) | 2 (2)
Gastro-intestinal bleed (Gastrointestinal disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
Hair Loss (Skin and subcutaneous tissue disorders) | 1 (1)
Hand inflammation (Immune system disorders) | 1 (1)
Hand lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (General disorders) | 6 (9)
Heart palpitations (Cardiac disorders) | 1 (2)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Hyperbilirubinemia (Hepatobiliary disorders) | 3 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (39)
Hyperkalemia (Renal and urinary disorders) | 8 (14)
Hypernatremia (Renal and urinary disorders) | 1 (1)
Hyperphosphatemia (Renal and urinary disorders) | 11 (22)
Hypertension (Cardiac disorders) | 7 (9)
Hyperuricema (Renal and urinary disorders) | 8 (16)
Hypoalbuminemia (Blood and lymphatic system disorders) | 4 (4)
Hypocalcemia (Renal and urinary disorders) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (8)
Hypokalemia (Renal and urinary disorders) | 3 (4)
Hyponatremia (Renal and urinary disorders) | 3 (7)
Hypophosphatemia (Renal and urinary disorders) | 9 (13)
Hypoxia (Cardiac disorders) | 1 (1)
Infected nose ulcer (Infections and infestations) | 1 (1)
Infusion reaction (Immune system disorders) | 1 (1)
Infusion-related reaction (Immune system disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)
Jaw discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Light-headedness (General disorders) | 1 (1)
Lymphocyte count increased (Blood and lymphatic system disorders) | 1 (1)
Mild bruising (Vascular disorders) | 1 (1)
Mouth sores (Skin and subcutaneous tissue disorders) | 2 (3)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 6 (7)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail Fragility (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6)
Neutropenia (Blood and lymphatic system disorders) | 18 (83)
Nose bleed (General disorders) | 3 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Paronychia in right toe (Infections and infestations) | 1 (2)
Petechia (Vascular disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prostate CA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rapid heart rate (Cardiac disorders) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 11 (16)
Rib pain (bruise) (Musculoskeletal and connective tissue disorders) | 2 (3)
Scalp inflammation (Skin and subcutaneous tissue disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Sinus tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin lesions (Skin and subcutaneous tissue disorders) | 1 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach pain (left side) (Gastrointestinal disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (128)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (3)
UTI (Renal and urinary disorders) | 1 (1)
Visual Change (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02315768/Prot_SAP_000.pdf